CLINICAL TRIAL: NCT00187330
Title: A Randomized Placebo Controlled Trial of Intravenous N-Acetylcysteine (NAC) As A Renal Protective Agent for Prevention of Renal Dysfunction Following Cardiopulmonary Bypass (CPB)
Brief Title: A Study of The Effectiveness of N-Acetylcysteine in Kidney Protection Following Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 724180589; R03-45; www.psifoundation.org
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-08

CONDITIONS: Heart Disease; Renal Insufficiency
Keywords: cardiopulmonary bypass; renal insufficiency; cardiac surgery; n-acetylcysteine
MeSH Terms: conditions — Heart Diseases; Renal Insufficiency

INTERVENTIONS:
Drug: Intravenous N-acetylcysteine

SUMMARY:
N-acetylcysteine is a medication that has most commonly been used in the past to prevent liver damage after an acetaminophen overdose. N-acetylcysteine has also been used in patients with pre-existing kidney damage to prevent further kidney damage resulting from dye that is used in tests such as angiograms (dye studies). This study hopes to prove that this medication may also help to protect kidneys from the damage caused by the heart-lung machine during cardiac surgery. This damage to the kidneys happens to patients undergoing cardiac surgery requiring the use of the heart-lung machine. Kidney failure after surgery is a serious complication (2-30% of patients with kidney problems can develop it) and it can lead to short term and long-term dialysis as well as death (there is up to a 30% death rate once kidney failure develops). The study will test if intravenous N-acetylcysteine is safe and effective in preventing kidney problems after cardiac surgery using the heart-lung machine. Approximately 104 patients will be enrolled at Sunnybrook and Women's College Health Science Centre. The study has been reviewed and approved by the ethics committee at Sunnybrook and Women's College Health Science Centre. The study will compare the effects of N-acetylcysteine with those of placebo (salt solution). The study medication (either N-acetylcysteine or placebo) will be given in addition to your usual medication and surgical procedures.

DETAILED DESCRIPTION:
Background:

N-acetylcysteine (NAC) is an oral or intravenous agent that replenishes glutathione which in turn allows for the formation of glutathione peroxidase, an important enzyme in the degradation cascade of reactive free oxygen radicals. NAC has been shown to reduce recurrent cardiac events in the setting of ischemic injury, and help prevent progression of renal dysfunction in patients with chronic renal failure exposed to nephrotoxic dye for radiographic studies. Cardiopulmonary bypass (CPB) has been shown be nephrotoxic that may be through the production of oxygen free radicals produced as a consequence of: a systemic inflammatory response to the pump, renal hypoperfusion and loss of pulsatile flow to the kidney during CPB. Renal dysfunction post cardiac surgery can lead to short or long term dialysis, and an increase in mortality rate. NAC therefore may be an ideal agent to preserve renal function in those patients who require exposure to CPB and are at high risk of developing postoperative renal dysfunction. The hypothesis tested in this study is that IV NAC may minimize postoperative renal dysfunction sustained by exposure to the cardiopulmonary bypass circuit.

Objectives:

This study will answer the question of whether perioperative intravenous N-Acetylcysteine (NAC) will be effective in reducing postoperative renal dysfunction as measured by a change peak creatinine from baseline values greater than or equal to 50μmol/L between placebo and NAC groups in adult, elective patients at high risk of renal insufficiency following exposure to cardiopulmonary bypass (CPB). This study is a randomized, placebo controlled, double blind trial that addresses the following objective:

1.To determine if intravenous N-Acetylcysteine (NAC) is effective in reducing post cardiopulmonary bypass renal dysfunction.

It is hypothesized that IV NAC will provide renal protection and may be an effective prophylactic option for patients at high risk of postoperative renal failure after exposure to CPB, and avoiding the ensuing high mortality rate associated with this.

Study Design:

This study will consist of a single centre, randomized, stratified, double blind, placebo controlled trial of intraoperative use of placebo or IV N-acetylcysteine (n=104 patients).

Study population:

Includes those patients with preoperative renal dysfunction (serum creatinine level 140 μmol/L or greater or a calculated glomerular filtration rate of 50 mL/min or less), or a risk factor score for postoperative renal dysfunction that adds up to 6 or more based on the following scale:

Score Risk Factor:

3 scheduled for redo cardiac surgery 3 scheduled for valve surgery 2 age greater than 69 at time of surgery 2 known diabetic (Type I or II) 2 congestive heart failure 2 treated hypertension 2 chronic obstructive pulmonary disease 2 preoperative stroke

1 left ventricular function -grade 3 or 4 (seen on echo or angiogram)

1 New York Heart Association Class 3 or 4

Exclusion Criteria:

Patient is participating in another trial

* Patient has received NAC in the past 48 hours.
* Patient has allergy to N-acetylcysteine.
* Patient scheduled for off-pump surgery or an extracardiac procedure (pericardiectomy etc.)
* Patient requires emergent surgery
* Patient scheduled for a procedure involving circulatory arrest.
* Patient requires chronic dialysis (peritoneal or hemodialysis)
* Patient unable to give informed consent (dementia, does not speak English, etc.)
* Patient has a recent history of cancer (in last five years) or untreated cancer

Randomization:

Patients will be randomized to either placebo or IV NAC (one to one allocation). There will be four strata. The four strata consist of the major divisions of isolated CABG surgery and valve surgery and the subdivisions of risk factor only patients, and patients with preoperative renal insufficiency. The patients will be randomized to each of these three strata using a permuted-block randomization with block sizes of 4. The randomization number will be kept by pharmacy personnel and be available for unblinding in case of any emergencies which would include anaphylaxis, hypotension (mean bp less than 60 mmHg), and liver failure. Blinding will be preserved as the IV NAC and placebo will be dispensed in identical IV solution bags that cannot be distinguished.

Intervention:

Patients will be randomized to receive either NAC (150 mg/kg bolus over 15 minutes after induction and 50 mg/kg/hr infusion during cardiopulmonary bypass) or placebo (same amount of saline both for bolus and infusion).

We also have provided standard guidelines suggested in the perioperative management of these patients as it pertains to renal protection including the use of co-interventions such as IV fluid management, pulsatile CPB, and use of vasopressors to maintain adequate perfusion pressures both during and following CPB.

Blinding:

The patients and caregivers will be blinded to the treatment group as the placebo will be identical to the IV NAC in appearance. The research personnel collecting data will also be blinded. The pharmacy personnel will be the only ones aware of the treatment assignments. Blinding will not be breached except for emergency situations as outlined above. The cardiac surgeon and anesthetist will be asked if they believe their patient is on study drug to ensure blinding has been preserved.

Intention to Treat:

The study will include those patients who do not tolerate NAC and do not receive the full NAC dosage because of adverse events in an intention to treat manner. These patients who have not have the full maneuver will therefore be included in the final analysis.

Outcomes:

The primary outcome that will be compared between NAC and placebo groups will be the increase in serum creatinine from preoperative baseline level after exposure to CPB. The secondary outcomes will include glomerular filtration rate (as calculated by serum creatinine, and demographic variables as well as serum cystatin C), blood urea nitrogen, early dialysis (in-hospital), in-hospital mortality, postoperative myocardial infarction (MI), peak troponin, stroke, and postoperative low output syndrome. Adverse events such as hypotension, anaphylaxis and alteration of coagulation parameters will be documented.

Implication of Potential Results:

If this study shows renal protection with IV NAC it could be used as an effective prophylactic option for patients at high risk of postoperative renal failure and the ensuing high mortality rate associated with this.

ELIGIBILITY:
Inclusion Criteria:

* The study includes those patients with preoperative renal dysfunction (serum creatinine level 140 μmol/L or greater or a calculated glomerular filtration rate of 50 mL/min or less), or a risk factor score for postoperative renal dysfunction that adds up to 6 or more based on the following scale:

Score Risk Factor:

* 3 scheduled for redo cardiac surgery
* 3 scheduled for valve surgery
* 2 age greater than 69 at time of surgery
* 2 known diabetic (Type I or II)
* 2 congestive heart failure
* 2 treated hypertension
* 2 chronic obstructive pulmonary disease
* 2 preoperative stroke
* 1 left ventricular function -grade 3 or 4 (seen on echo or angiogram)
* 1 New York Heart Association Class 3 or 4

Exclusion Criteria:

* Patient is participating in another trial
* Patient has received NAC in the past 48 hours.
* Patient has allergy to N-acetylcysteine.
* Patient scheduled for off-pump surgery or an extracardiac procedure (pericardiectomy etc.)
* Patient requires emergent surgery
* Patient scheduled for a procedure involving circulatory arrest.
* Patient requires chronic dialysis (peritoneal or hemodialysis)
* Patient unable to give informed consent (dementia, does not speak English, etc.)
* Patient has a recent history of cancer (in last five years) or untreated cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104
Dates: Start 2004-03; Study Completion 2005-08

PRIMARY OUTCOMES:
The change in serum creatinine between NAC and placebo groups from preoperative baseline levels to peak postoperative levels after exposure to CPB.

SECONDARY OUTCOMES:
Include change in GFR, BUN and troponin; early dialysis; in-hospital mortality; postop MI; stroke; and postop LOS. SNPs related to renal insufficiency, ischemia, and inflammation will be analyzed in relation to serum inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Guru, MD, Principal Investigator — University of Toronto, Sunnybrook and Women's College Health Sciences Centre; Stephen E Fremes, MD, Study Chair — Sunnybrook Health Sciences Centre